CLINICAL TRIAL: NCT01517243
Title: Alternating Targeted Therapy in Patients With Metastatic Renal Cell Carcinoma: A Phase II Study of Alternating Sunitinib and Temsirolimus
Brief Title: Phase II Study of Alternating Sunitinib and Temsirolimus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Lionel.D.Lewis, MD, Medical Director of the Dartmouth Clinical Trials Office, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1011
Record Dates: First submitted 2012-01-17; First posted 2012-01-25 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Metastatic Renal Cell Carcinoma; sunitinib; alternating; temsirolimus
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alternating Sunitinib and Temsirolimus (Experimental): A cycle is defined as:
  Sunitinib 50mg by mouth daily for 4 weeks followed by a two week rest Temsirolimus 25mg IV weekly for 4 weeks followed by a two week rest
  Interventions: Drug: Sunitinib; Drug: Temsirolimus

INTERVENTIONS:
Drug: Sunitinib — Sunitinib 50mg by mouth daily for 4 weeks followed by a two week rest
  Other Names: Sutent
Drug: Temsirolimus — Temsirolimus 25mg IV weekly for 4 weeks followed by a two week rest
  Other Names: TORISEL®

SUMMARY:
In the past 5 years, treatment for metastatic Renal Cell Carcinoma (mRCC) has focused on agents directed at blocking tumor and vascular growth pathways. Sunitinib blocks the vascular endothelial growth factor receptor (VEGFr) and temsirolimus is an inhibitor of mammalian target of rapamycin (mTOR). Both sunitinib and temsirolimus are FDA approved agents for mRCC. When agents like these are given together, the toxicity increases but they can be given safely, at full doses, sequentially. We hypothesize that alternating these agents will double the progression free survival (PFS) of the agents when given sequentially.

DETAILED DESCRIPTION:
SUMMARY: Alternating Targeted Therapy in Patients with Metastatic Renal Cell Carcinoma: A Phase II Study of Alternating Sunitinib and Temsirolimus

Patients with measurable metastatic renal cell carcinoma (any histology) are eligible. All patients will be treated as outlined below with sunitinib alternating with temsirolimus.

Patients will be treated continuously, until evidence of progression of disease, or for up to two cycles following disappearance of all disease.

A cycle is defined as:

Sunitinib 50mg by mouth daily for 4 weeks followed by a two week rest Temsirolimus 25mg IV weekly for 4 weeks followed by a two week rest

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed metastatic renal cell cancer with evaluable disease.
* Patients must be at least 2 weeks from their last immunotherapy, surgery or chemotherapy (6 weeks for nitrosureas) and recovered from all ill effects.
* Karnofsky Performance Status ≥60%
* Life expectancy ≥ twelve weeks
* Adequate end organ function:

Cardiac Left ventricular ejection fraction (LVEF) ≥lower limit of institutional normal (LLN) as assessed by echocardiography (ECHO) . The same modality used at baseline must be applied for subsequent evaluations.

* Women should not be lactating and, if of childbearing age, have a negative pregnancy test within two weeks of entry to the study and practicing acceptable forms of birth control
* Appropriate Contraception in both sexes
* The patient must be competent and signed informed consent.

EXCLUSION CRITERIA

* Concomitant second malignancy except for non-melanoma skin cancer, and non-invasive cancer such as cervical CIS, superficial bladder cancer without local recurrence, breast CIS.
* In patients with a prior history of invasive malignancy, less than five years in complete remission.
* Have evidence of significant co-morbid illness such as uncontrolled diabetes, hypertension or active infection that would preclude treatment on this regimen.
* Prior treatment with either sunitinib or temsirolimus
* Clinically significant gastrointestinal abnormalities
* Presence of uncontrolled infection.
* Prolongation of corrected QT interval (QTc) > 480 milliseconds - History of any one or more of the following cardiovascular conditions within the past 12 months:

  1. Cardiac angioplasty or stenting
  2. Myocardial infarction
  3. Unstable angina
  4. Coronary artery by-pass graft surgery
  5. Symptomatic peripheral vascular disease
  6. Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* History of cerebrovascular accident (CVA) including transient ischemic attack (TIA) within the past 12 months.
* History of pulmonary embolism or untreated deep venous thrombosis (DVT)within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anticoagulating agents for at least 6 weeks are eligible.
* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of

  ≥150 or diastolic blood pressure (DBP) of ≥ 90. Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry.
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
* Evidence of active bleeding or bleeding diathesis
* Hemoptysis within 6 weeks of first dose of study drug.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
* Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study.
* Is now undergoing and/or has undergone in the 14 days immediately prior to first dose of study drug any minor surgeries (i.e. skin biopsy, tooth extraction, etc.) and recovered from all ill effects.
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to sunitinib or temsirolimus.
* Untreated brain metastasis. (Brain metastases that are stable based on radiographic evidence 4 weeks after radiation and/or surgery are permitted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-09-22 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lionel D Lewis, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- United States (2):
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Vermont, Vermont Cancer Center, Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 37 participants signed consent, of those, 3 withdrew consent and 15 were screen failures
Groups:
- Alternating Sunitinib and Temsirolimus: A cycle is defined as:
  Sunitinib 50mg by mouth daily for 4 weeks followed by a two week rest Temsirolimus 25mg IV weekly for 4 weeks followed by a two week rest
  Sunitinib: Sunitinib 50mg by mouth daily for 4 weeks followed by a two week rest
  Temsirolimus: Temsirolimus 25mg IV weekly for 4 weeks followed by a two week rest
Period: Overall Study
Arm/Group | Alternating Sunitinib and Temsirolimus
Started | 19 (Defined as those participants that signed consent and started treatment)
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Number of Participants Classified by Tumor Histology/Cytology: A cycle is defined as:
  Sunitinib 50mg by mouth daily for 4 weeks followed by a two week rest Temsirolimus 25mg IV weekly for 4 weeks followed by a two week rest
  Sunitinib: Sunitinib 50mg by mouth daily for 4 weeks followed by a two week rest
  Temsirolimus: Temsirolimus 25mg IV weekly for 4 weeks followed by a two week rest
Arm/Group | Number of Participants Classified by Tumor Histology/Cytology
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19
Tumor Histology/Cytology [Number; unit: participants]
  Clear Cell | 16
  Papillary | 1
  Unclassified | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: To determine the time to disease progression in metastatic renal cell carcinoma patients treated with alternating targeted therapy. This time interval constitutes the metric progression free survival time.
Time Frame: From the date of randomization until the first documented disease progression or date of death from any cause, evaluated every 12 weeks throughout duration of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Alternating Sunitinib and Temsirolimus
Number analyzed (Participants) | 19
Months | 8.8 [6.8 to 25.2]

2. Secondary Outcome: Clinical Response Rate as Measured by Best Response Achieved
Description: To be assigned a status of partial response or complete response, changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 4 weeks after the criteria for response are first met. In the case of stable disease, follow-up measurements must have met the stable disease criteria at least once after study entry at a minimum interval (in general, not less than 6-8 weeks) that is defined in the study protocol. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Every 12 weeks from randomization until progression, estimated time frame is 18 months
Measure: Number; unit: Participants
Arm/Group | Alternating Sunitinib and Temsirolimus
Number analyzed (Participants) | 19
Participants
  Partial Response | 5
  Stable Disease | 9
  Progression of Disease | 3
  Not Evaluable | 2

3. Secondary Outcome: To Characterize the Toxicity Profile
Description: The toxicity profile will be characterized by observations of AEs and SAEs graded by the CTCAE criteria v4.0.
Time Frame: Throughout the duration of the patient remaining on study treatment which was a median time of 8 months
Measure: Number; unit: participants
Arm/Group | Alternating Sunitinib and Temsirolimus
Number analyzed (Participants) | 19
participants | 19

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time consent was obtained until 4 weeks post progression, approximately 10 months
Arm/Group | Alternating Sunitinib and Temsirolimus
All-Cause Mortality (participants affected / at risk) | 1/19
Serious Adverse Events (participants affected / at risk) | 4/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alternating Sunitinib and Temsirolimus (N=19)
Dysarthia (Nervous system disorders) | 1 (1)
Ischemia Cerebrovascular (stroke) (Vascular disorders) | 1 (1)
Muscle Weakness- right sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Urosepsis (Renal and urinary disorders) | 1 (1)
Pneumonia (w/ sepsis) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alternating Sunitinib and Temsirolimus (N=19)
Hypertension (Cardiac disorders) | 5 (6)
Alanine aminotransferase increased (Investigations) | 3 (4)
Alkaline phosphatase increased (Investigations) | 3 (4)
Allergic reaction (rash) (Immune system disorders) | 6 (7)
Amylase increased (Investigations) | 3 (6)
Anemia (Investigations) | 9 (9)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 2 (4)
Cholesterol high (Investigations) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2)
Concentration impairment (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Creatinine increased (Investigations) | 8 (12)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (10)
Dizziness (Nervous system disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Dysesthesia (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Ear Pain (Ear and labyrinth disorders) | 2 (2)
Edema Limbs (General disorders) | 4 (9)
Edema Face (General disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Facial Muscle Weakness (Nervous system disorders) | 1 (1)
Facial pain (General disorders) | 2 (2)
Fatigue (General disorders) | 14 (17)
Fever (General disorders) | 4 (4)
Flu like symptoms (General disorders) | 1 (1)
Spinal Fracture (C6) (Injury, poisoning and procedural complications) | 1 (1)
Fracture (rib) (Injury, poisoning and procedural complications) | 1 (1)
Gastronintestinal pain (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hair color changes (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (6)
Hearing Impaired (Ear and labyrinth disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (7)
Hypotension (Cardiac disorders) | 1 (1)
Hypothyroidism (Metabolism and nutrition disorders) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Infusion site extravasation (General disorders) | 1 (2)
INR increased (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Pain- joint (General disorders) | 2 (2)
Blood Lactate dehydrogenase increased (Investigations) | 1 (1)
Wound complication- hernia (Injury, poisoning and procedural complications) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Lip Infection (Infections and infestations) | 2 (3)
Lipase Increased (Investigations) | 3 (4)
Lung infection (Infections and infestations) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 10 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 (8)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3)
Phlebitis (Vascular disorders) | 2 (2)
Platelet count decreased (Investigations) | 6 (10)
White blood cell decreased (Investigations) | 3 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Proteinuria (Renal and urinary disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 3 (4)
Pain- right iliac (General disorders) | 1 (1)
Libido increased (Psychiatric disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2)
urinary tract infection (Infections and infestations) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (3)
Watering eyes (Eye disorders) | 1 (1)
Weight loss (Investigations) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT01517243/Prot_SAP_000.pdf